CLINICAL TRIAL: NCT03857321
Title: Device Study for Intranasal Delivery of Insulin
Brief Title: Study of Nasal Insulin to Fight Forgetfulness - Device Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00055429
Record Dates: First submitted 2019-02-22; First posted 2019-02-27 (Actual); Results first posted 2025-08-20 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2024-12

CONDITIONS: Mild Cognitive Impairment; Cognitive Impairment
Keywords: Intranasal Delivery of Insulin; Cognitive Testing; Nasal Insulin
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Insulin

STUDY DESIGN:
Intervention Model Description: At study entry, participants will be randomized to receive either an acute dose of insulin or of placebo first and the other substance on a second visit.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Neither participants or site personnel will know whether insulin or saline is being administered. Exceptions will be the study nurse who is directly involved in preparing the insulin or placebo, as well as preparing DSMB reports.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Insulin first, then placebo (Experimental): Participants will be randomly assigned to receive regular insulin (U100, 20 IU) administered with an intranasal nebulizer-like device. Participants in this arm will then receive placebo at visit 3 during second intervention period.
  Interventions: Drug: Insulin; Other: Placebo; Device: intranasal nebulizer-like device
- Placebo first, then insulin (Experimental): Participants will be randomly assigned to receive placebo administered with an intranasal nebulizer-like device. At visit 3 during second intervention period, participants in this arm will receive insulin.
  Interventions: Drug: Insulin; Other: Placebo; Device: intranasal nebulizer-like device

INTERVENTIONS:
Drug: Insulin — 20 IU Humulin® R U-100 (NDC: 0002-8215, Eli Lilly & Company)
  Other Names: Humulin® R U-100
Other: Placebo — Matching placebo (sterile saline) to 20 IU Humulin® R U-100
  Other Names: placebo to Humulin® R U-100; Sterile saline
Device: intranasal nebulizer-like device — Participants will be assigned to receive placebo or regular insulin (U100, 20 IU) administered through an intranasal nebulizer-like device.

SUMMARY:
The SNIFF Device study will involve using a device to administer insulin through each participant's nose or intra-nasally. Insulin is a hormone that is produced in the body. It works by lowering levels of glucose (sugar) in the blood. This study is measuring how much insulin the device delivers. In addition, this study will look at the effects of insulin or placebo administered intra-nasally using a nebulizer-like device on memory, blood, and cerebral spinal fluid.

DETAILED DESCRIPTION:
The aim of this study is to determine the ability of an intranasal delivery device to increase levels of insulin in cerebrospinal fluid (CSF).

A growing body of evidence suggests that insulin plays a role in normal memory processes and that insulin abnormalities may contribute to cognitive and brain changes associated with Alzheimer's disease (AD). Interestingly, insulin administered to the nasal cavity is transported within a few minutes into the brain, but does not affect blood sugar or insulin levels.

The study will consist of a single site, randomized, double-blind trial comparing the acute effects of INI (20 International Units) or placebo delivered with nebulizer-like device on CSF insulin levels, AD biomarkers and memory. At study entry, participants will be randomized to receive either an acute dose of insulin or placebo first, and the other substance on a second visit. Participants who are cognitively normal or who have aMCI (n=30) will be enrolled. The primary outcome measure will be to test the hypothesis that CSF insulin levels will increase 30 minutes after receiving a 20 International Units dose of insulin delivered with a nebulizer-like device, compared to levels achieved 30 minutes after placebo.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English
* Cognitively normal or diagnosis of aMCI
* Stable medical condition for 3 months prior to screening visit
* Stable medications for 4 weeks prior to the screening and study visits
* Clinical laboratory values must be within normal limits or, if abnormal, must be judged to be clinically insignificant by the study physician

Exclusion Criteria:

* A diagnosis of dementia
* History of a clinically significant stroke
* Current evidence or history in past two years of epilepsy, head injury with loss of consciousness, any major psychiatric disorder including psychosis, major depression, bipolar disorder
* Diabetes (type I or type II) insulin dependent and non-insulin dependent diabetes mellitus
* Current or past use of insulin or any other anti-diabetic medication within 5 years of Screening visit.
* History of cancer five years prior to screening (history of skin melanoma or stable prostate cancer are not exclusionary)
* History of seizure within past five years
* Pregnancy or possible pregnancy.
* Use of anticoagulants warfarin (Coumadin) and dabigatran (Pradaxa)
* Residence in a skilled nursing facility at screening
* Use of an investigational agent within two months of screening visit
* Regular use of alcohol, narcotics, anticonvulsants, antiparkinsonian medications, or any other exclusionary medications

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Craft, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albert MS, DeKosky ST, Dickson D, Dubois B, Feldman HH, Fox NC, Gamst A, Holtzman DM, Jagust WJ, Petersen RC, Snyder PJ, Carrillo MC, Thies B, Phelps CH. The diagnosis of mild cognitive impairment due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):270-9. doi: 10.1016/j.jalz.2011.03.008. Epub 2011 Apr 21. PMID 21514249
- [Background] Baker H, Spencer RF. Transneuronal transport of peroxidase-conjugated wheat germ agglutinin (WGA-HRP) from the olfactory epithelium to the brain of the adult rat. Exp Brain Res. 1986;63(3):461-73. doi: 10.1007/BF00237470. PMID 3758265
- [Background] Baker LD, Cross DJ, Minoshima S, Belongia D, Watson GS, Craft S. Insulin resistance and Alzheimer-like reductions in regional cerebral glucose metabolism for cognitively normal adults with prediabetes or early type 2 diabetes. Arch Neurol. 2011 Jan;68(1):51-7. doi: 10.1001/archneurol.2010.225. Epub 2010 Sep 13. PMID 20837822
- [Background] Balin BJ, Broadwell RD, Salcman M, el-Kalliny M. Avenues for entry of peripherally administered protein to the central nervous system in mouse, rat, and squirrel monkey. J Comp Neurol. 1986 Sep 8;251(2):260-80. doi: 10.1002/cne.902510209. PMID 3782501
- [Background] Benedict C, Hallschmid M, Hatke A, Schultes B, Fehm HL, Born J, Kern W. Intranasal insulin improves memory in humans. Psychoneuroendocrinology. 2004 Nov;29(10):1326-34. doi: 10.1016/j.psyneuen.2004.04.003. PMID 15288712
- [Background] Benedict C, Kern W, Schultes B, Born J, Hallschmid M. Differential sensitivity of men and women to anorexigenic and memory-improving effects of intranasal insulin. J Clin Endocrinol Metab. 2008 Apr;93(4):1339-44. doi: 10.1210/jc.2007-2606. Epub 2008 Jan 29. PMID 18230654
- [Background] Bodian, D. and H. A. Howe (1941).
- [Background] Born J, Lange T, Kern W, McGregor GP, Bickel U, Fehm HL. Sniffing neuropeptides: a transnasal approach to the human brain. Nat Neurosci. 2002 Jun;5(6):514-6. doi: 10.1038/nn849. No abstract available. PMID 11992114
- [Background] Broadwell RD, Balin BJ. Endocytic and exocytic pathways of the neuronal secretory process and trans-synaptic transfer of wheat germ agglutinin-horseradish peroxidase in vivo. J Comp Neurol. 1985 Dec 22;242(4):632-50. doi: 10.1002/cne.902420410. PMID 2418083
- [Background] Cavanna AE, Trimble MR. The precuneus: a review of its functional anatomy and behavioural correlates. Brain. 2006 Mar;129(Pt 3):564-83. doi: 10.1093/brain/awl004. Epub 2006 Jan 6. PMID 16399806
- [Background] Chiu SL, Chen CM, Cline HT. Insulin receptor signaling regulates synapse number, dendritic plasticity, and circuit function in vivo. Neuron. 2008 Jun 12;58(5):708-19. doi: 10.1016/j.neuron.2008.04.014. PMID 18549783
- [Background] Craft S, Baker LD, Montine TJ, Minoshima S, Watson GS, Claxton A, Arbuckle M, Callaghan M, Tsai E, Plymate SR, Green PS, Leverenz J, Cross D, Gerton B. Intranasal insulin therapy for Alzheimer disease and amnestic mild cognitive impairment: a pilot clinical trial. Arch Neurol. 2012 Jan;69(1):29-38. doi: 10.1001/archneurol.2011.233. Epub 2011 Sep 12. PMID 21911655
- [Background] Craft S, Peskind E, Schwartz MW, Schellenberg GD, Raskind M, Porte D Jr. Cerebrospinal fluid and plasma insulin levels in Alzheimer's disease: relationship to severity of dementia and apolipoprotein E genotype. Neurology. 1998 Jan;50(1):164-8. doi: 10.1212/wnl.50.1.164. PMID 9443474
- [Background] Craft S, Watson GS. Insulin and neurodegenerative disease: shared and specific mechanisms. Lancet Neurol. 2004 Mar;3(3):169-78. doi: 10.1016/S1474-4422(04)00681-7. PMID 14980532
- [Background] De Felice FG, Vieira MN, Bomfim TR, Decker H, Velasco PT, Lambert MP, Viola KL, Zhao WQ, Ferreira ST, Klein WL. Protection of synapses against Alzheimer's-linked toxins: insulin signaling prevents the pathogenic binding of Abeta oligomers. Proc Natl Acad Sci U S A. 2009 Feb 10;106(6):1971-6. doi: 10.1073/pnas.0809158106. Epub 2009 Feb 2. PMID 19188609
- [Background] Faber, H. K. (1938).
- [Background] Fairbrother, R. W. and E. W. Hurst (1930).
- [Background] Fishel MA, Watson GS, Montine TJ, Wang Q, Green PS, Kulstad JJ, Cook DG, Peskind ER, Baker LD, Goldgaber D, Nie W, Asthana S, Plymate SR, Schwartz MW, Craft S. Hyperinsulinemia provokes synchronous increases in central inflammation and beta-amyloid in normal adults. Arch Neurol. 2005 Oct;62(10):1539-44. doi: 10.1001/archneur.62.10.noc50112. PMID 16216936
- [Background] Francis GJ, Martinez JA, Liu WQ, Xu K, Ayer A, Fine J, Tuor UI, Glazner G, Hanson LR, Frey WH 2nd, Toth C. Intranasal insulin prevents cognitive decline, cerebral atrophy and white matter changes in murine type I diabetic encephalopathy. Brain. 2008 Dec;131(Pt 12):3311-34. doi: 10.1093/brain/awn288. Epub 2008 Nov 16. PMID 19015157 (Retraction: PMID 24860127 Brain. 2014 Jun;137(Pt 6):e283)
- [Background] Frolich L, Blum-Degen D, Bernstein HG, Engelsberger S, Humrich J, Laufer S, Muschner D, Thalheimer A, Turk A, Hoyer S, Zochling R, Boissl KW, Jellinger K, Riederer P. Brain insulin and insulin receptors in aging and sporadic Alzheimer's disease. J Neural Transm (Vienna). 1998;105(4-5):423-38. doi: 10.1007/s007020050068. PMID 9720972
- [Background] Galasko D, Bennett D, Sano M, Ernesto C, Thomas R, Grundman M, Ferris S. An inventory to assess activities of daily living for clinical trials in Alzheimer's disease. The Alzheimer's Disease Cooperative Study. Alzheimer Dis Assoc Disord. 1997;11 Suppl 2:S33-9. PMID 9236950
- [Background] Gasparini L, Gouras GK, Wang R, Gross RS, Beal MF, Greengard P, Xu H. Stimulation of beta-amyloid precursor protein trafficking by insulin reduces intraneuronal beta-amyloid and requires mitogen-activated protein kinase signaling. J Neurosci. 2001 Apr 15;21(8):2561-70. doi: 10.1523/JNEUROSCI.21-08-02561.2001. PMID 11306609
- [Background] Gil-Bea FJ, Solas M, Solomon A, Mugueta C, Winblad B, Kivipelto M, Ramirez MJ, Cedazo-Minguez A. Insulin levels are decreased in the cerebrospinal fluid of women with prodomal Alzheimer's disease. J Alzheimers Dis. 2010;22(2):405-13. doi: 10.3233/JAD-2010-100795. PMID 20847404
- [Background] Hallschmid M, Benedict C, Schultes B, Born J, Kern W. Obese men respond to cognitive but not to catabolic brain insulin signaling. Int J Obes (Lond). 2008 Feb;32(2):275-82. doi: 10.1038/sj.ijo.0803722. Epub 2007 Sep 11. PMID 17848936
- [Background] Hong M, Lee VM. Insulin and insulin-like growth factor-1 regulate tau phosphorylation in cultured human neurons. J Biol Chem. 1997 Aug 1;272(31):19547-53. doi: 10.1074/jbc.272.31.19547. PMID 9235959
- [Background] Hughes CP, Berg L, Danziger WL, Coben LA, Martin RL. A new clinical scale for the staging of dementia. Br J Psychiatry. 1982 Jun;140:566-72. doi: 10.1192/bjp.140.6.566. PMID 7104545
- [Background] Illum L. Nasal drug delivery: new developments and strategies. Drug Discov Today. 2002 Dec 1;7(23):1184-9. doi: 10.1016/s1359-6446(02)02529-1. PMID 12547019
- [Background] Kern W, Born J, Schreiber H, Fehm HL. Central nervous system effects of intranasally administered insulin during euglycemia in men. Diabetes. 1999 Mar;48(3):557-63. doi: 10.2337/diabetes.48.3.557. PMID 10078556
- [Background] Kristensson K, Olsson Y. Uptake of exogenous proteins in mouse olfactory cells. Acta Neuropathol. 1971;19(2):145-54. doi: 10.1007/BF00688493. No abstract available. PMID 5126829
- [Background] Kupila A, Sipila J, Keskinen P, Simell T, Knip M, Pulkki K, Simell O. Intranasally administered insulin intended for prevention of type 1 diabetes--a safety study in healthy adults. Diabetes Metab Res Rev. 2003 Sep-Oct;19(5):415-20. doi: 10.1002/dmrr.397. PMID 12951650
- [Background] Lee CC, Kuo YM, Huang CC, Hsu KS. Insulin rescues amyloid beta-induced impairment of hippocampal long-term potentiation. Neurobiol Aging. 2009 Mar;30(3):377-87. doi: 10.1016/j.neurobiolaging.2007.06.014. Epub 2007 Aug 10. PMID 17692997
- [Background] Minoshima S, Frey KA, Foster NL, Kuhl DE. Preserved pontine glucose metabolism in Alzheimer disease: a reference region for functional brain image (PET) analysis. J Comput Assist Tomogr. 1995 Jul-Aug;19(4):541-7. doi: 10.1097/00004728-199507000-00006. PMID 7622680
- [Background] Minoshima S, Koeppe RA, Frey KA, Kuhl DE. Anatomic standardization: linear scaling and nonlinear warping of functional brain images. J Nucl Med. 1994 Sep;35(9):1528-37. PMID 8071705
- [Background] Morris JC, Ernesto C, Schafer K, Coats M, Leon S, Sano M, Thal LJ, Woodbury P. Clinical dementia rating training and reliability in multicenter studies: the Alzheimer's Disease Cooperative Study experience. Neurology. 1997 Jun;48(6):1508-10. doi: 10.1212/wnl.48.6.1508. PMID 9191756
- [Background] Petersen RC, Doody R, Kurz A, Mohs RC, Morris JC, Rabins PV, Ritchie K, Rossor M, Thal L, Winblad B. Current concepts in mild cognitive impairment. Arch Neurol. 2001 Dec;58(12):1985-92. doi: 10.1001/archneur.58.12.1985. PMID 11735772
- [Background] Pontiroli AE, Alberetto M, Secchi A, Dossi G, Bosi I, Pozza G. Insulin given intranasally induces hypoglycaemia in normal and diabetic subjects. Br Med J (Clin Res Ed). 1982 Jan 30;284(6312):303-6. doi: 10.1136/bmj.284.6312.303. PMID 6800439
- [Background] Reger MA, Watson GS, Frey WH 2nd, Baker LD, Cholerton B, Keeling ML, Belongia DA, Fishel MA, Plymate SR, Schellenberg GD, Cherrier MM, Craft S. Effects of intranasal insulin on cognition in memory-impaired older adults: modulation by APOE genotype. Neurobiol Aging. 2006 Mar;27(3):451-8. doi: 10.1016/j.neurobiolaging.2005.03.016. Epub 2005 Jun 16. PMID 15964100
- [Background] Reger MA, Watson GS, Green PS, Baker LD, Cholerton B, Fishel MA, Plymate SR, Cherrier MM, Schellenberg GD, Frey WH 2nd, Craft S. Intranasal insulin administration dose-dependently modulates verbal memory and plasma amyloid-beta in memory-impaired older adults. J Alzheimers Dis. 2008 Apr;13(3):323-31. doi: 10.3233/jad-2008-13309. PMID 18430999
- [Background] Reger MA, Watson GS, Green PS, Wilkinson CW, Baker LD, Cholerton B, Fishel MA, Plymate SR, Breitner JC, DeGroodt W, Mehta P, Craft S. Intranasal insulin improves cognition and modulates beta-amyloid in early AD. Neurology. 2008 Feb 5;70(6):440-8. doi: 10.1212/01.WNL.0000265401.62434.36. Epub 2007 Oct 17. PMID 17942819
- [Background] Rivera EJ, Goldin A, Fulmer N, Tavares R, Wands JR, de la Monte SM. Insulin and insulin-like growth factor expression and function deteriorate with progression of Alzheimer's disease: link to brain reductions in acetylcholine. J Alzheimers Dis. 2005 Dec;8(3):247-68. doi: 10.3233/jad-2005-8304. PMID 16340083
- [Background] Rubin, D. B. (1987). Multiple Imputation for Nonresponse in Surveys. Hoboken, New Jersey, John Wiley & Sons, Inc
- [Background] Sakane T, Akizuki M, Taki Y, Yamashita S, Sezaki H, Nadai T. Direct drug transport from the rat nasal cavity to the cerebrospinal fluid: the relation to the molecular weight of drugs. J Pharm Pharmacol. 1995 May;47(5):379-81. doi: 10.1111/j.2042-7158.1995.tb05814.x. PMID 7494186
- [Background] Sano M, Raman R, Emond J, Thomas RG, Petersen R, Schneider LS, Aisen PS. Adding delayed recall to the Alzheimer Disease Assessment Scale is useful in studies of mild cognitive impairment but not Alzheimer disease. Alzheimer Dis Assoc Disord. 2011 Apr-Jun;25(2):122-7. doi: 10.1097/WAD.0b013e3181f883b7. PMID 20921876
- [Background] Selkoe DJ. Soluble oligomers of the amyloid beta-protein impair synaptic plasticity and behavior. Behav Brain Res. 2008 Sep 1;192(1):106-13. doi: 10.1016/j.bbr.2008.02.016. Epub 2008 Feb 17. PMID 18359102
- [Background] Shipley MT. Transport of molecules from nose to brain: transneuronal anterograde and retrograde labeling in the rat olfactory system by wheat germ agglutinin-horseradish peroxidase applied to the nasal epithelium. Brain Res Bull. 1985 Aug;15(2):129-42. doi: 10.1016/0361-9230(85)90129-7. PMID 3840049
- [Background] Stockhorst U, de Fries D, Steingrueber HJ, Scherbaum WA. Insulin and the CNS: effects on food intake, memory, and endocrine parameters and the role of intranasal insulin administration in humans. Physiol Behav. 2004 Oct 30;83(1):47-54. doi: 10.1016/j.physbeh.2004.07.022. PMID 15501490
- [Background] Thorne RG, Emory CR, Ala TA, Frey WH 2nd. Quantitative analysis of the olfactory pathway for drug delivery to the brain. Brain Res. 1995 Sep 18;692(1-2):278-82. doi: 10.1016/0006-8993(95)00637-6. PMID 8548316
- [Background] Thorne RG, Pronk GJ, Padmanabhan V, Frey WH 2nd. Delivery of insulin-like growth factor-I to the rat brain and spinal cord along olfactory and trigeminal pathways following intranasal administration. Neuroscience. 2004;127(2):481-96. doi: 10.1016/j.neuroscience.2004.05.029. PMID 15262337
- [Background] Townsend M, Mehta T, Selkoe DJ. Soluble Abeta inhibits specific signal transduction cascades common to the insulin receptor pathway. J Biol Chem. 2007 Nov 16;282(46):33305-33312. doi: 10.1074/jbc.M610390200. Epub 2007 Sep 13. PMID 17855343
- [Background] Weiss P, Holland Y. Neuronal dynamics and axonal flow, ii. The olfactory nerve as model test object. Proc Natl Acad Sci U S A. 1967 Feb;57(2):258-64. doi: 10.1073/pnas.57.2.258. No abstract available. PMID 16591462
- [Background] Worsley KJ, Evans AC, Marrett S, Neelin P. A three-dimensional statistical analysis for CBF activation studies in human brain. J Cereb Blood Flow Metab. 1992 Nov;12(6):900-18. doi: 10.1038/jcbfm.1992.127. PMID 1400644
- [Background] Zhao L, Teter B, Morihara T, Lim GP, Ambegaokar SS, Ubeda OJ, Frautschy SA, Cole GM. Insulin-degrading enzyme as a downstream target of insulin receptor signaling cascade: implications for Alzheimer's disease intervention. J Neurosci. 2004 Dec 8;24(49):11120-6. doi: 10.1523/JNEUROSCI.2860-04.2004. PMID 15590928
- [Background] Zhao WQ, Townsend M. Insulin resistance and amyloidogenesis as common molecular foundation for type 2 diabetes and Alzheimer's disease. Biochim Biophys Acta. 2009 May;1792(5):482-96. doi: 10.1016/j.bbadis.2008.10.014. Epub 2008 Nov 5. PMID 19026743

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The insulin-placebo/placebo-insulin sequence is a critical component of the study. It was counterbalanced in order to address potential practice effects for the Auditory-Verbal Learning Test (AVLT).
Groups:
- Insulin First, Then Placebo; Placebo First, Then Insulin: Participants in one group will receive regular insulin administered with an intranasal nebulizer-like device and will crossover to placebo for the second half of the trial. Participants in the other group will receive placebo first and crossover to insulin for the second half of the trail. Crossover occurs at visit 3.
  The insulin-placebo/placebo-insulin sequence is a critical component of the study. It was counterbalanced in order to address potential practice effects for the Auditory-Verbal Learning Test (AVLT). It is well known that memory test scores are lower the first time the test is taken, and then are higher the second time. The phenomenon is known as the practice effect. They are higher the second time because participants have been exposed to the memory stimuli previously. Thus if placebo is always administered first and insulin second, it may appear that the memory scores have improved due to the insulin, when the improvement is due instead to practice effects.
  Insulin: 20 IU Humulin® R U-100 (NDC: 0002-8215, Eli Lilly & Company)
  Placebo: Matching placebo (sterile saline) to 20 IU Humulin® R U-100
Period: Overall Study
Arm/Group | Insulin First, Then Placebo | Placebo First, Then Insulin
Started | 11 | 9
Completed | 11 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Participants in one group will receive regular insulin administered with an intranasal nebulizer-like device and will crossover to placebo for the second half of the trial. Participants in the other group will receive placebo first and crossover to insulin for the second half of the trail. Crossover occurs at visit 3. Insulin: 20 IU Humulin® R U-100 (NDC: 0002-8215, Eli Lilly & Company) Placebo: Matching placebo (sterile saline) to 20 IU Humulin® R U-100
Arm/Group | All Participants
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 67.8 [62 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: CSF Insulin Levels
Description: Levels of insulin in cerebrospinal fluid after being delivered with the device. This will help to determine the ability of an intranasal delivery device to increase levels of insulin in cerebrospinal fluid (CSF)
Time Frame: 30 minutes after intervention administration
Population: The insulin-placebo/placebo-insulin sequence is a critical component of the study. The order was counterbalanced to address a phenomenon known as Practice Effect when giving the AVLT. When memory test are given a second time scores are higher because participants have been exposed to the memory stimuli previously. Thus if placebo is always given first and insulin second, it may appear that the memory scores have improved due to the insulin when the improvement is due instead to Practice Effects.
Measure: Mean (Full Range); unit: microUnits/mL
Arm/Group | Insulin First, Then Placebo | Placebo First, Then Insulin
Number analyzed (Participants) | 11 | 9
microUnits/mL
  First Intervention: number analyzed (Participants) | 11 | 0
  First Intervention | 0.14 [0.01 to 0.26] |
  Second Intervention: number analyzed (Participants) | 0 | 9
  Second Intervention |  | 0.15 [0.06 to 0.40]

2. Secondary Outcome: The Auditory-Verbal Learning Test (AVLT)
Description: memory measure in which participant hears a list of 12 words over 3 trials, and is asked to recall them immediately after hearing them, then again after a 45 minute delay. Total possible score is 36 for immediate recall and 12 for delayed recall. Higher scores are better.
Time Frame: 5 minutes before lumbar puncture, and immediately following lumbar puncture
Population: as for outcome 1
Measure: Mean (Full Range); unit: average words recalled
Arm/Group | Insulin First, Then Placebo | Placebo First, Then Insulin
Number analyzed (Participants) | 10 | 9
average words recalled
  First Intervention 5 minutes before lumbar puncture: number analyzed (Participants) | 10 | 0
  First Intervention 5 minutes before lumbar puncture | 7.1 [4.6 to 10.4] |
  First Intervention Immediately following lumbar puncture: number analyzed (Participants) | 10 | 0
  First Intervention Immediately following lumbar puncture | 4.9 [0 to 9] |
  Second Intervention 5 minutes before lumbar puncture: number analyzed (Participants) | 0 | 9
  Second Intervention 5 minutes before lumbar puncture |  | 9.4 [5.2 to 11.6]
  Second Intervention Immediately following lumbar puncture: number analyzed (Participants) | 0 | 9
  Second Intervention Immediately following lumbar puncture |  | 8.9 [3 to 14]

3. Secondary Outcome: CSF Levels of AB42
Description: Levels of the 42 amino acid isoform of the beta amyloid peptide
Time Frame: 30 minutes after intervention administration
Population: as for outcome 1
Measure: Mean (Full Range); unit: pg/ml
Arm/Group | Insulin First, Then Placebo | Placebo First, Then Insulin
Number analyzed (Participants) | 11 | 9
pg/ml
  Insulin first, then placebo: number analyzed (Participants) | 11 | 0
  Insulin first, then placebo | 524.5 [207.0 to 1086.5] |
  Placebo first, then insulin: number analyzed (Participants) | 0 | 9
  Placebo first, then insulin |  | 536 [244.0 to 757.5]

4. Secondary Outcome: CSF Levels of Total Tau
Description: Levels of the tau protein
Time Frame: 30 minutes after intervention administration
Population: as for outcome 1
Measure: Mean (Full Range); unit: pg/ml
Arm/Group | Insulin First, Then Placebo | Placebo First, Then Insulin
Number analyzed (Participants) | 11 | 9
pg/ml
  Insulin first, then placebo: number analyzed (Participants) | 11 | 0
  Insulin first, then placebo | 431.4 [126.0 to 880.5] |
  Placebo first, then insulin: number analyzed (Participants) | 0 | 9
  Placebo first, then insulin |  | 267.3 [125.5 to 687.0]

5. Secondary Outcome: CSF Levels Phospho-tau 181
Description: Levels of the tau phosphorylated at isotope 181
Time Frame: 30 minutes after intervention administration
Population: as for outcome 1
Measure: Mean (Full Range); unit: pg/ml
Arm/Group | Insulin First, Then Placebo | Placebo First, Then Insulin
Number analyzed (Participants) | 11 | 9
pg/ml
  Insulin first, then placebo: number analyzed (Participants) | 11 | 0
  Insulin first, then placebo | 61.5 [21.0 to 107.3] |
  Placebo first, then insulin: number analyzed (Participants) | 0 | 9
  Placebo first, then insulin |  | 40.6 [20.4 to 109.0]

ADVERSE EVENTS:
Time Frame: Up to Week 6
Groups:
- Insulin: Participants will be randomly assigned to receive regular insulin (U100, 20 IU) administered with an intranasal nebulizer-like device.
  Insulin: 20 IU Humulin® R U-100 (NDC: 0002-8215, Eli Lilly & Company)
  intranasal nebulizer-like device: Participants will be assigned to receive placebo or regular insulin (U100, 20 IU) administered through an intranasal nebulizer-like device.
- Placebo: Participants will be randomly assigned to receive placebo administered with an intranasal nebulizer-like device.
  Placebo: Matching placebo (sterile saline) to 20 IU Humulin® R U-100
  intranasal nebulizer-like device: Participants will be assigned to receive placebo or regular insulin (U100, 20 IU) administered through an intranasal nebulizer-like device.
Arm/Group | Insulin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 4/20 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin (N=20) | Placebo (N=20)
vasovagal episode (Nervous system disorders) | 1 (1) | 0 (0)
low back discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
tired (General disorders) | 1 (1) | 0 (0)
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-07): https://cdn.clinicaltrials.gov/large-docs/21/NCT03857321/Prot_SAP_002.pdf
  • Informed Consent Form (2023-09-20): https://cdn.clinicaltrials.gov/large-docs/21/NCT03857321/ICF_001.pdf